CLINICAL TRIAL: NCT03010826
Title: Pharmacological Recruitment of Endogenous Neural Precursors to Promote Pediatric White Matter Repair: Establishing Correlations Between Visual Outcomes, Saccadic Function and MEG Oscillations in Children With Demyelinating Disorders in Comparison to Healthy Control Children
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, E. Ann Yeh, Associate Scientist, Research Institute, The Hospital for Sick Children
Other Study IDs: 1000053920
Record Dates: First submitted 2017-01-03; First posted 2017-01-05 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Demyelinating Disease
MeSH Terms: conditions — Demyelinating Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 40 Demyelinating Disease patients
- 40 Non-patient participants

SUMMARY:
The neural circuits in our brains require a layer of insulation in order to transmit signals in a rapid and efficient fashion. This insulation is called White Matter and is comprised of a specific type of brain cell called an oligodendrocytes. Damage to brain white matter occurs following injury and in disorders like Multiple Sclerosis and results in sensory, motor, and cognitive problems. Currently there are no effective medical therapies to promote brain repair and reduce disability following damage to white matter. In this project, we hope to change the situation by encouraging the brain itself to generate new oligodendrocytes and thus new white matter. Our first step is to find measures sensitive to white matter growth.

ELIGIBILITY:
Inclusion Criteria:

* Experienced a demyelinating event (Only applicable to patient subjects)
* Between the ages of 5 years to 18 years and 11 months of age
* Has either English as his or her native language or has had at least two years of schooling in English

Exclusion Criteria:

* Children with non-demyelinating etiologies of white matter dysfunction (i.e., metabolic disorders, vasculitis, and non-specific MRI abnormalities
* Is younger than 5 years of age
* Is 18 years and 11 of age or older
* Has a prior history of traumatic brain injury, neurological disorder, cerebral palsy, developmental delay, or learning disability
* Requires sedation for brain scanning
* Is claustrophobic, as brain scanning requires children to enter a tunnel in the MRI machine

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: There will be a total of 80 participants in this study. The study population consists of both patients (demyelinating disease) and non-patient participants (healthy volunteers).
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2016-12; Primary Completion 2018-11-16 (Actual); Study Completion 2018-11-16 (Actual)

PRIMARY OUTCOMES:
Neuronal responses during pro/anti-saccade eye movements | 60 minutes
  Video-based eye tracking monocularly in the MEG and binocularly outside the MEG
Electrical potentials initiated by brief visual stimuli | 10 minutes
  Visual Evoked Potentials (VEP)
MRI scans of the brain, including Diffusion Tensor Imagine (DTI) | 90 minutes
Neurocognitive Testing | 90 minutes
  Computerized Penn Neurocognitive Battery
High contrast visual acuity | 10 minutes
Low contrast visual acuity; colour vision; visual fields testing; OCT testing; | 10 minutes
Colour vision testing | 10 minutes
Visual fields testing | 20 minutes
Optical coherence tomography (OCT) | 25 minutes
Neurological Exam - Standard physical exam performed by neurologist to determine the Expanded Disability Status Scale (EDSS) score. | 20 minutes
Clinical Interview | 10 minutes

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Queen's University, Kingston, Ontario
  - Hospital for Sick Children, Toronto, Ontario